CLINICAL TRIAL: NCT03618173
Title: Efficiency of IV Dexamethasone Compared to Placebo, Administrated After a Lower Limb Blockade is Done, on the Post Operative Pain in Children : a Controled, Randomised, Double Blind Study
Brief Title: Efficiency of IV Dexamethasone, Administered After a Lower Limb Blockade, on the Post Operative Pain in Children
Acronym: DEXPED
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-000314-38
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: IV Drug Usage
Keywords: dexamethasone; analgesia; lower limb blockade; children; pediatric
MeSH Terms: conditions — Agnosia | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexamethasone (Experimental): IV dexamethasone group : dexamethasone administrated at the induction of general anesthesia, at the dose of 0,2mg/kg (= 0,2mL/kg of a syringe with a 1mg/mL concentration) maximum 8mg (=8mL).
  Interventions: Drug: Dexamethasone
- Placebos (Placebo Comparator): IV placebo group : saline serum is administrated at the induction of general anesthesia, at the dose of 0,2mL/kg, maximum 8mL.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dexamethasone — IV dexamethasone at the dose of 0,2mg/kg = 0,2mL/kg of a solution of 1mg/mL max 8mg
  Other Names: IV dexamethasone
  Arms: dexamethasone
Drug: Placebos — IV saline serum at the dose of 0,2mL/kg maximum 8mL
  Other Names: IV saline serum
  Arms: Placebos

SUMMARY:
Intravenous dexamethasone (IV) can be used alone in adults as an adjunct to peri-nerves blocks, for diffusion blocks.

In pediatrics, dexamethasone is used daily according to the assessment of the anesthetist, by extension of the recommendations of the adult, as adjuvant in perinervous blocks although no study has been published yet concerning his interest. However, the physiology of the child is not superimposable to that of the adult (renal function, volume of distribution, plasma protein binding ...).

We thus wish to study the effectiveness of the administration of IV dexamethasone at the time of anesthetic induction in the prolongation of the duration of the block of the lower limbs in the child and its repercussion on the postoperative consumption of morphine.

Main Objective : Evaluate the efficiency, compared to placebo, of IV dexamethasone at the dose of 0.2 mg / kg administered as a bolus at the time of anesthetic induction, on the early postoperative pain (first 24 hours) in the child of 6 to 15 years undergoing surgery that requires the achievement of a peri-neural block of the lower limb after general anesthesia

Secondary objectives :

* Evaluate the efficiency of 0,2mg/kg IV dexamathasone administrated at anesthesia induction compared to placebo, on the increase of the delay of first post operative morphinic consumption in children from 6 to 15 who are qualified for a lower limb surgery with a loco-regional anesthesia.
* Evaluate that 0,2mg/kg IV dexamathasone administrated at anesthesia induction compared to placebo, doesn't increase the lower limb motor blokade duration in children from 6 to 15 who are qualified for a lower limb surgery with a loco-regional anesthesia
* Evaluate the efficiency of 0,2mg/kg IV dexamathasone administrated at anesthesia induction compared to placebo, on the decrease of post operative nausea and vomiting in children from 6 to 15 who are qualified for a lower limb surgery with a loco-regional anesthesia

Principal endpoint :

-Morphinic consumption in the post operative 24H

Secondary endpoints :

* delay between the realisation of the lower limb blockade ans the first - consumption of morphinic
* duration the the motor blockade
* prevalence of post opérative nausea/vomiting

DETAILED DESCRIPTION:
Time 1: Pre-anesthetic consultation

Recruitment is performed during the pre-anesthetic consultation, between D-90 and D-2 of the date of operation. The eligibility criteria will be checked and if the child is eligible to participate in the study, oral and written information about the study is given to the child's parents (or, failing that, to their legal representatives) by the anesthetist doctor. Minors will receive information adapted to their ability to understand. It can not be overridden by the refusal of the child or the revocation of his acceptance. The investigator will give the parents the consent form The parents then have a minimum of 48 hours to decide whether to participate in the study of their child.

In all cases, an anesthesiologist doctor will be reachable (through the secretariat) at any time in case of additional questions during the reflection period.

Time n ° 2: Pre-anesthetic visit

If the parents and the child agree to participate in this study and after a new eligibility check, the consent signed by both parents will be collected the day before the intervention during the pre-anesthetic visit.

The randomization will then be carried out and two groups will be created:

* A first group receiving 0.2 mg / kg of IV dexamethasone at the time of anesthetic induction
* A second group receiving the same volume of placebo (physiological saline)

The anesthetist will send to the pharmacy, on a prescription, the results of the randomization (assignment code) the day before the procedure.

The drugs in the study will be prepared by the pharmacy department of the University Hospital of Nancy at most 21 days in advance of the intervention. Indeed, a syringe for each randomization list (stratification on algebra level) will always be planned in advance and ready to be used for inclusion early in the morning (between 7:30 and 9:30).

The packaging will be identical to guarantee the double blind. The pharmacy will send the drug to the operating room on the morning of the operation via a specific drug transport.

On the morning of the operation, all patients included will receive a premedication with midazolam 0.3mg / kg per os 30 minutes max 10mg before surgery.

The patient is then asleep (general anesthesia) according to the protocols in force (initial induction by inhaled sevoflurane and then peripheral venous route (VVP) and injection of sufentanil 0.1 gamma / kg and propofol 2-3mg / kg or VVP pose then IV anesthesia directly in the larger ones).

Then a block of the lower limb with 0.3mL / kg of ropivacaine at the concentration of 2mg / mL, ultrasound guided with or without neurostimulation is performed.

The patient then receives according to his group:

* either 0.2 mg / kg of IV dexamethasone at the time of anesthetic induction
* or the same volume of placebo (physiological saline) at the time of anesthetic induction.

Maintenance of general anesthesia is done by sevoflurane with sufentanil reinjection at the discretion of the anesthesiologist.

In the intraoperative period, the patient will receive a systematic injection of paracetamol 15mg / kg IVL 30 minutes before the end of the surgical procedure.

Once the operation is complete, the patient is transferred to the post-interventional surveillance room with awakening and evaluation of the pain (by EVA scale) and postoperative nausea (by questioning the child), noting the hours of statement. The existence of a motor block of the operated lower limb is also evaluated and recorded. Thereafter, the patient returns to conventional service with regular evaluation (every 4 hours) of pain and nausea / vomiting (every 4 hours).

The pain intensity will be evaluated by a scale validated from the age of 6: evaluation by analogue verbal scale (EVA) giving a painful intensity over 100: 100/100 being the maximum intensity imaginable, 0/100 the absence of pain.

The occurrence of postoperative nausea and vomiting will be assessed as follows: no nausea / vomiting, nausea without vomiting, nausea and vomiting.

If the EVA is greater than 30 in the 24 hours postoperative: an injection of Nalbuphine 0.2mg / kg IVL or morphine 0.1mg / kg max 3mg every 4 to 6 hours will be performed; in the event of failure (persistence of an EVA> 30 to 30 mins), a new dose of paracetamol 15mg / kg may be administered again 6 hours after the first dose injected intraoperatively.

In the event of nausea and / or postoperative vomiting, ondansetron 0.1mg / kg every 8h will be administered and then in case of failure at 30 minutes, droperidol 10 microgram / kg every 8h.

ELIGIBILITY:
Inclusion Criteria:

* Children from 6 to 15 who are qualified for a lower limb surgery with a loco-regional anesthesia with an anesthesic consultation between 90 to 2 days before the surgery
* Legal guardian agreement
* Children who are affiliated to the social security
* Information of minor subjects adapted to their ability to understand

Exclusion Criteria:

* Children who presents a contraindication to the single shot IV dexamethasone
* Septic surgery
* Diabetes
* Corticoid treatment in the 7 days before the surgery - outpatient surgery
* Handicapped or impaired children
* Pregnant patient
* Peri-nerval catheter
* Children who are privated from their liberty because of a court or administrative decision or need psychiatric care
* Uncontrolled psychotic state
* Pregnant patients

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Morphinic consumption in the post operative 24H | within 24 hours after dexamethasone or saline serum administration
  total morphinic consumption in morphine equivalent in mg

SECONDARY OUTCOMES:
Delay between the realisation of the lower limb blockade ans the first - consumption of morphinic | within 24 hours after dexamethasone or saline serum administration
  delay in minutes between the realization of the lower limb blockade and the first consumption of morphinic
Duration the the motor blockade | within 24 hours after dexamethasone or saline serum administration
  motor blockade evaluated with the bromide score over 6 points, duration to recover a score of 6/6 (no more blockade) in minutes
Prevalence of post opérative nausea/vomiting | within 24 hours after dexamethasone or saline serum administration
  evaluated with no nausea/vomiting, nausea OR vomiting, nausea AND vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Claude Meistelman, Principal Investigator — University Professor in CHRU Nancy

REFERENCES:
- [Derived] Vautrin N, Thilly N, Bernard Y, Wurtz F, Meistelman C. Protocol of DEXPED trial: efficacy of intravenous dexamethasone, administered at the time of analgesic blocking of the lower limb, on postoperative pain in children: a randomised, placebo-controlled, double-blind trial. BMJ Open. 2020 Sep 30;10(9):e036863. doi: 10.1136/bmjopen-2020-036863. PMID 32998920